CLINICAL TRIAL: NCT06745466
Title: Disentangling the Effects of Daily Stress, Sleep, and Sex Hormones on Accelerated Vascular Aging in Midlife Women
Acronym: V-RISES
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2207199; R21AG090810 (NIH)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Estrogen; Premenopause
Keywords: Premenopause; Estrogen; Stress; Sleep; Vascular function
MeSH Terms: interventions — ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Natural cycle (No Intervention): Participants will undergo study measurements during the follicular phase of their natural menstrual cycle.
- No to Low Endogenous Estrogen (Experimental): Participants will undergo study measurements during 10 days of daily ganirelix acetate (Antagon) injections.
  Interventions: Drug: ganirelix acetate

INTERVENTIONS:
Drug: ganirelix acetate — Ganirelix acetate (Antagon) will be used to prevent endogenous production of ovarian hormones in young women. Ganirelix is derived from native GnRH, and acts by competitively blocking GnRH receptors on the pituitary and subsequent pathways. Thus, administration of the GnRH antagonist (GnRHant) suppresses steroidogenesis, leading to low or undetectable serum estrogen and progesterone concentrations, which occurs within two days of initiation of administration. Women will self-administer subcutaneous injections (0.25 mg/day in 0.5 ml of normal saline) of the GnRH antagonist ganirelix acetate (Antagon, Organon, Inc., West Orange, New Jersey,) every day for ~12-15 days (starting on day ~2-4 of the menstrual cycle). Testing will occur on day 3-4 and day14-15 of using Antagon.
  Other Names: Antagon
  Arms: No to Low Endogenous Estrogen

SUMMARY:
The purpose of this study is to identify the impact of estradiol (E2) on the associations between (a) responsivity to daily stress or (b) sleep variability with vascular function in midlife premenopausal women.

DETAILED DESCRIPTION:
In the last 20 years, deaths due to cardiovascular disease (CVD) have increased by up to 30% in midlife women. This increase in CVD risk in midlife women is at least partially explained by the declines in estradiol (E2) that occur across the menopausal transition. This loss of E2 induces vascular dysfunction, a major contributor to increased CVD risk. Nevertheless, we have shown that declines in vascular function are evident in some midlife premenopausal women, suggesting that vascular dysfunction-associated CVD risk cannot solely be explained by the loss of E2. Emerging factors that may help explain vascular dysfunction in midlife women include greater emotional vulnerability to daily stressors and poorer sleep health. However, not yet know is the extent to which daily stress and sleep health independently impact vascular function in midlife premenopausal women or the degree to which these associations are influenced by E2. The objective of this project is to test the central hypothesis that (a) greater negative affective responsivity to daily stressors and (b) greater sleep variability will each be related to more severe declines in vascular function in midlife premenopausal women and that these associations will be magnified during E2 suppression (simulated menopause) compared to the follicular phase of the menstrual cycle/placebo phase of hormonal contraception. We will assess affective responsitivy to daily stressors and device-measured sleep characteristics for 10 consecutive days and cutaneous microvascular endothelial function before and during pharmacological E2 suppression.

The investigators will assess multiple dynamic aspects of daily stress processes for 10 consecutive days (mobile app). Investigators will concurrently objectively assess sleep variability (ActiGraph wGT3X). Immediately before and after completion of these ambulatory assessments, Investigators will assess microvascular endothelial function using intradermal microdialysis coupled with laser Doppler flowmetry. Participants will complete two 10-day measurement bursts:The first will occur during the follicular phase of their menstrual cycle or the low hormone/placebo phase of hormonal contraception; The second will occur during supression of endogenous ovarian hormone production via GnRH antagonist ganirelix acetate.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 40-55
* Premenopausal

Exclusion Criteria:

* Pregnancy (including a positive urine pregnancy test), planning to become pregnant, or breast-feeding
* Peri- or post-menopausal
* Unstable or diagnosed chronic clinical disease, including cardiovascular, metabolic, renal, hepatic, autonomic, autoimmune, or dermatological disease
* Current or lifetime major psychiatric illness (e.g., major depressive disorder, bipolar disorder, schizophrenia, eating disorders)
* History of hysterectomy (complete or partial), polycystic ovary syndrome, endometrial hyperplasia, irregular menstrual cycles, or endometrial ablation
* Suspected potential presence of obstructive sleep apnea (STOP-Bang score >3) or insomnia (Insomnia Severity Index score >15)
* Current or recent (within 8 wks) use of medications that could conceivably alter cardiovascular function or sleep health
* Changes or alterations in medication status (starting a new, additional, or different medication or changing the dose of a current medication)
* Body mass index >35 kg/m2
* Tobacco or nicotine use, including vaping and electronic cigarettes
* Working night-time or rotating shift work within the previous 3 months
* Trans-meridian travel during study enrollment (inclusive of the entire duration of enrollment and the period between testing cycles)
* Known allergies to pharmacological agents/drugs
* Current use of long-acting reversible contraception (LARC; e.g., IUDs, birth control implants)
* Known latex allergy

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Endothelium-dependent dilation (EDD) | Immediately before and after each 10-day measurement burst
  EDD will be calculated as the area under the dose-response curve (AUC) to ascending concentrations of acetylcholine.
Negative affective response to daily stressors | 10-day measurement burst
  Within-person composite slope between daily stressors and daily negative affect
Sleep variability | 10-day measurement burst
  Sleep onset standard deviation (minutes) estimated via actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Jody Greaney, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No